CLINICAL TRIAL: NCT01530893
Title: Are the Cardiovascular Responses of Individuals at Mild to Moderate Cardiovascular Risk Influenced by Dietary Flavonoid Sub-class and Dietary Form?
Brief Title: Flavonoids, Blood Pressure and Blood Vessel Function
Acronym: FASTCHECK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of East Anglia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Basic Science
Other Study IDs: FASTCHECK
Record Dates: First submitted 2012-02-01; First posted 2012-02-10 (Estimated); Last update posted 2014-02-28 (Estimated); Status verified 2014-02

CONDITIONS: Cardiovascular Disease Risk Reduction
Keywords: flavonoids; vascular function; randomised controlled trial; placebo controlled

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Intervention group A: flavanones (Experimental): All experimental days will be exactly the same. All volunteers will attend the clinical research and trial unit in a fasted state. Prior to test administration, baseline vascular function will be assessed and biological samples taken by a trained and qualified research nurse. Subsequently, assessments will be repeated at times corresponding to anticipated peak plasma concentration of the flavonoid of interest.
  Interventions: Dietary Supplement: Flavanone - supplement; Other: Flavanone - food; Other: Flavanone - placebo
- Intervention group B: isoflavones (Experimental): All experimental days will be exactly the same. All volunteers will attend the clinical research and trial unit in a fasted state. Prior to test administration, baseline vascular function will be assessed and biological samples taken by a trained and qualified research nurse. Subsequently, assessments will be repeated at times corresponding to anticipated peak plasma concentration of the flavonoid of interest.
  Interventions: Dietary Supplement: Isoflavone - supplement; Other: Isoflavone - food; Other: Isoflavone - placebo; Dietary Supplement: Isoflavone - metabolite supplement
- Intervention group C: Flavan-3-ols (Experimental): All experimental days will be exactly the same. All volunteers will attend the clinical research and trial unit in a fasted state. Prior to test administration, baseline vascular function will be assessed and biological samples taken by a trained and qualified research nurse. Subsequently, assessments will be repeated at times corresponding to anticipated peak plasma concentration of the flavonoid of interest.
  Interventions: Dietary Supplement: Flavan-3-ol - supplement; Other: Flavan-3-ol - food; Other: Flavan-3-ol - placebo
- Intervention group D: Anthocyanins (Experimental): All experimental days will be exactly the same. All volunteers will attend the clinical research and trial unit in a fasted state. Prior to test administration, baseline vascular function will be assessed and biological samples taken by a trained and qualified research nurse. Subsequently, assessments will be repeated at times corresponding to anticipated peak plasma concentration of the flavonoid of interest.
  Interventions: Dietary Supplement: Anthocyanin - supplement; Other: Anthocyanin - food; Other: Anthocyanin - placebo

INTERVENTIONS:
Dietary Supplement: Flavanone - supplement — acute single optimal dose
  Arms: Intervention group A: flavanones
Other: Flavanone - food — acute single dose
  Arms: Intervention group A: flavanones
Other: Flavanone - placebo — acute single dose (flavanone free)
  Arms: Intervention group A: flavanones
Dietary Supplement: Isoflavone - supplement — acute single optimal dose
  Arms: Intervention group B: isoflavones
Other: Isoflavone - food — acute single optimal dose
  Arms: Intervention group B: isoflavones
Other: Isoflavone - placebo — acute single dose (isoflavone free)
  Arms: Intervention group B: isoflavones
Dietary Supplement: Isoflavone - metabolite supplement — acute single optimal dose of commercial product
  Arms: Intervention group B: isoflavones
Dietary Supplement: Flavan-3-ol - supplement — acute single optimal dose
  Arms: Intervention group C: Flavan-3-ols
Other: Flavan-3-ol - food — acute single optimal dose
  Arms: Intervention group C: Flavan-3-ols
Other: Flavan-3-ol - placebo — acute single dose (flavan-3-ol free)
  Arms: Intervention group C: Flavan-3-ols
Dietary Supplement: Anthocyanin - supplement — acute single optimal dose
  Arms: Intervention group D: Anthocyanins
Other: Anthocyanin - food — acute single optimal dose
  Arms: Intervention group D: Anthocyanins
Other: Anthocyanin - placebo — acute single dose (anthocyanin free)
  Arms: Intervention group D: Anthocyanins

SUMMARY:
The primary aim of this placebo-controlled study is to determine whether flavonoids beneficially affect markers of cardiovascular disease risk in healthy subjects at elevated cardiovascular risk.

The underlying mechanisms of action of flavonoids will be assessed on blood biomarkers and we will assess the effects of the food matrix, and aspects of isoflavone metabolism.

DETAILED DESCRIPTION:
The study population will be healthy males (aged 50-75 years) at elevated risk of cardiovascular (CV) disease.

A target of 60 participants will be required to complete the study and a total of 70 subjects will be targeted (n=70 subjects * ~85% anticipated completion rate = 60 subjects to complete the study).

This placebo-controlled study will test the relative efficacy of 4 different flavonoid sub-classes ((i) flavan-3-ol, (ii) anthocyanin, (iii) flavanone and (iv) isoflavone).

Accordingly, subjects will be randomised to one of the four flavonoid study groups ((i) to (iv) outlined above), and then will consume each of the following treatments in random order:

1. dietary flavonoid + placebo supplement
2. placebo food + commercially available/produced flavonoid supplement
3. placebo food + placebo supplement

Additionally, an isoflavone metabolite will be fed to establish potential vascular effects.

Each sub-class will be assessed separately and a 1 week wash-out period between treatments will be observed.

At each assessment visit, vascular function will be assessed pre- and post-intervention, with subsequent assessments made to coincide with anticipated peak plasma concentrations.

Dietary intake will be monitored during the study and participants will be required to adhere to a range of dietary and lifestyle restrictions within 3 days of each assessment to reduce potential confounding of the data assessment of interest.

A standard battery of vascular function tests will be performed on all intervention groups, with each assessment visit performed in an identical manner.

ELIGIBILITY:
Inclusion Criteria:

* Males
* 50 to 75 years old
* At elevated risk of CV disease
* Screening blood pressure of < 160/90mmHg (at rest)
* Successful biochemical, haematological and urinalysis assessment at screening (as judged by clinical advisor)

Exclusion Criteria:

* Current smokers, or ex-smokers ceasing < 3 months ago
* Subjects with existing or significant past medical history of vascular disease or medical conditions likely to affect the study measures (as judged by clinical advisor)
* Those with known allergies to the intervention treatments
* Those unprepared to adhere to dietary restrictions during the trial
* Parallel participation in another research project which involves concurrent dietary intervention and/or sampling of biological fluids/material
* Having vaccinations (excluding the flu vaccination) or antibiotics within 3 months of start of trial, and those with vaccinations scheduled for during the trial
* Taking flavonoid containing food / dietary supplements likely to affect the study results
* Prescribed lipid lowering, hypertension, vasodilators (e.g. Viagra) or antibiotic medication
* Unsatisfactory biochemical, haematological or urinary assessment at screening, indicating abnormal; renal or liver function, full blood profile, impaired glucose handling, deranged lipids or measurements considered to be counter indicative of the study by the clinical advisor

Ages: 50 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2012-02; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in blood vessel control (pressure and endothelial function) at time points coinciding with postprandial [anticipated] peak plasma flavonoid concentration. | acute postprandial; up to 24 hours, dependent on flavonoid sub-classification studied
  Assessment of vascular function

SECONDARY OUTCOMES:
Differences in effects of flavonoids introduced by food matrix | acute postprandial; up to 24 hours dependent on flavonoid sub-classification studied

CONTACTS AND LOCATIONS:
Overall Officials: Aedin Cassidy, PhD, Principal Investigator — University of East Anglia
Locations (1):
- Department of Nutrition, Norwich Medical School, Norwich, Norfolk, United Kingdom

REFERENCES:
- [Derived] Hazim S, Curtis PJ, Schar MY, Ostertag LM, Kay CD, Minihane AM, Cassidy A. Acute benefits of the microbial-derived isoflavone metabolite equol on arterial stiffness in men prospectively recruited according to equol producer phenotype: a double-blind randomized controlled trial. Am J Clin Nutr. 2016 Mar;103(3):694-702. doi: 10.3945/ajcn.115.125690. Epub 2016 Feb 3. PMID 26843154
- [Derived] Schar MY, Curtis PJ, Hazim S, Ostertag LM, Kay CD, Potter JF, Cassidy A. Orange juice-derived flavanone and phenolic metabolites do not acutely affect cardiovascular risk biomarkers: a randomized, placebo-controlled, crossover trial in men at moderate risk of cardiovascular disease. Am J Clin Nutr. 2015 May;101(5):931-8. doi: 10.3945/ajcn.114.104364. Epub 2015 Mar 18. PMID 25788001